CLINICAL TRIAL: NCT00516308
Title: A Non-Randomized Study of the NightHawk Peripheral Plaque Excision System During Plaque Excision of Peripheral Arterial Disease
Acronym: NightHawk
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Other
Sponsor: FoxHollow Technologies (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FHT-P-07-004
Record Dates: First submitted 2007-08-13; First posted 2007-08-15 (Estimated); Last update posted 2008-01-18 (Estimated); Status verified 2008-01

CONDITIONS: Peripheral Vascular Diseases
Keywords: CLI; Critical Limb Ischemia; PAD; Paripheral Arterial Disease; Artherosclerosis; Leg pain; Cardiovascular; Atherectomy; NightHawk
MeSH Terms: conditions — Peripheral Vascular Diseases; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: NightHawk

SUMMARY:
To assess the proximity of the catheter to the vessel wall and to correlate excised tissue with images collected by the integrated Optical coherence Tomography (OCT) imaging system. The primary endpoints are correlation between OCT images and histological characterization of excised tissue.

ELIGIBILITY:
Inclusion Criteria:

1. Patient requires treatment for peripheral arterial disease (PAD).
2. Patient is willing and able to provide Informed Consent.
3. Patient has at least one focal, de novo infrainguinal lesion in a native vessel.
4. The minimum reference vessel diameter is 2.0 - 4.5 mm, dependent on the NightHawk device used.
5. The lesion is ≥ 50% stenosed by quantitative vascular angiography.
6. The lesion is ≤ 7 cm in length.
7. The patient must be able to take at least one form of anti-platelet or anti-thrombotic therapy.

Exclusion Criteria:

1. Patient presents with degree of limb disease or a co-existing medical condition that makes revascularization inappropriate.
2. The patient has diffuse peripheral arterial disease and/or the disease is heavily calcified.
3. Patient presents with concomitant disease contraindicating an endovascular intervention.
4. Patient is pregnant.
5. The patient has a hypersensitivity to contrast materials that cannot be adequately pretreated.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-08; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Austin Heart, Austin, Texas, United States